CLINICAL TRIAL: NCT03039894
Title: Improving School Engagement Among Early Adolescents: Evaluation of a Team-based Social Network Intervention
Brief Title: Grade Book Game Evaluation Among 6th Grade Students
Acronym: GG
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mitchell Wong, MD, PhD, Professor of Medicine; Faculty Mentor, University of California, Los Angeles
Other Study IDs: IRB#16-001059
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Adolescent Behaviors
Keywords: school-based, evaluation, interrupted time series
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: The middle school selected 2 advisory classrooms to participate in the Gradebook game during 6th grade. Students in these 2 classrooms were block randomized to teams by baseline grade book and student engagement scores. These small student teams stay together for an entire year and meet once or twice a week. Teams are led by 8th grade student team captains, picked by school staff for their positive leadership skills. Every 2 weeks throughout the year, teams are randomly matched in head-to-head competition. In each 2-week-long game (i.e. Gradebook Game), individual team members accrue points from teachers and administrators for academic performance, effort, and school behavior. Team wins are announced and public scoreboards are updated frequently. The investigators will collect student survey data at baseline and after the intervention, approximately 5-6 months apart.
  Interventions: Other: Gradebook Game
- Control: The middle school has chosen three 6th grade classrooms that will not play the Gradebook game. The investigators will collect school gradebook and behavior information weekly for 8 to 10 time points before and after the intervention is implemented. Students will complete a survey at baseline and after the intervention, approximately 5-6 months apart.

INTERVENTIONS:
Other: Gradebook Game — Students in the intervention group will spend time meeting as teams to review their scorecards, and do team-building activities, all of which will occur during non-content periods at school (Advisory and Enrichment).
  Groups: Intervention

SUMMARY:
School engagement is associated with children's long-term health and success. Students who are engaged in school have better academic outcomes and lower rates of risky health behaviors. The investigators partnered with Alliance College-Ready Middle Academy 12 (Alliance 12), a charter school in Los Angeles, to develop the "gradebook game", an intervention that aims to improve academic achievement, peer support, and school engagement. The game involves frequent feedback on students' school performance, team-based competition aligned with the school mission, and peer mentorship by team captains. For the 2016-2017 academic year, the investigators will assist Alliance 12 in implementing the gradebook game in two of its five 6th grade homerooms. The investigators plan to evaluate whether the game, as hypothesized, is effective in increasing school engagement, including academic performance and positive behavior.

In order to conduct this evaluation, the investigators plan to enroll 6th grade students by obtaining parental consent and student assent at the beginning of the school year. Students will be enrolled for the entire 2016-2017 academic year. All study procedures except for parental recruitment will occur during the school day. Participation in the study involves completing 2 student surveys and permitting the collection and analysis of student data from the online gradebook and behavior system. The investigators plan to use an interrupted time series design that will analyze student gradebook and behavior data at multiple time points before and after the game starts. The surveys will be completed at the beginning and end of the study period. Surveys will include measures of self-reported school engagement, age, gender, race/ethnicity, primary language at home, social and emotional well-being, social status, and peer support. Surveys will be administered via iPad.

If the pilot study demonstrates that the gradebook game is effective in promoting school engagement and academic achievement, it is anticipated that it could be widely adopted and more rigorously evaluated in a larger study. Because the gradebook game is a low-resource intervention, it could easily and sustainably be replicated, providing a much-needed tool for schools with low engagement.

DETAILED DESCRIPTION:
School engagement is critical to students' long-term success and appears to be strongly influenced by peer relationships. School engagement results from the interaction of the individual with the school context and is a multi-dimensional concept involving behavioral, emotional, and cognitive components. These include attendance, conduct, effort, participation, emotions towards school, identification with school, interest, and psychological investment in learning. Children who are engaged in school have higher levels of academic achievement and increased likelihood of occupational success as adults, even beyond that predicted by achievement. Children who are successful in school are also healthier adults, which is due in part to health risk behaviors that begin in adolescence. School engagement appears to protect against substance use and delinquency. Factors that have been associated with low levels of engagement (or disengagement) include trauma, stress, discrimination, and bullying, whereas supportive relationships with parents, peers, and teachers promote school engagement. Because school engagement is modifiable, it is an obvious target for school-based intervention.

Prior studies have documented interventions that improve school engagement, but effect sizes are generally small and they are resource-intensive and therefore difficult to implement widely. As far as the investigators know, none have used a social network or team-based behavioral economics approach. A partnership between UCLA and Alliance College-Ready Middle Academy #12 (Alliance 12), a charter middle school in Los Angeles led to the development of the novel Gradebook Game. This intervention aims to induce supportive social pressure aligned with a school's mission in order to promote school engagement and achievement. Sixth grade students are organized into teams by Advisory period and mentored by 8th grade team captains. Throughout the regular school day, students are assigned points for effort, achievement, and citizenship (as captured by the online gradebook and behavior tracker), which then get repackaged into weekly team scorecards for the Game. Teams compete against each other for total points in bi-weekly match-ups, and wins are rewarded with incentives tailored to the school's needs. This intervention is unique in bringing a team-based behavioral economics approach to impact school engagement. It is grounded in principles from two successful interventions: the Good Behavior Game and Peer Connection. The Gradebook Game Intervention has been piloted for feasibility in one Advisory group of 6th grade students at Alliance 12 during the Spring of 2016. If effective, it could feasibly be implemented widely and has the potential to transform social norms and school culture, providing a much-needed tool among schools with low student engagement.

The investigators plan to study the effectiveness of the Gradebook Game in promoting school engagement and achievement. This study would likely be the first to evaluate an intervention that utilizes team competition to generate social pressure and peer support around behaviors that promote success in school. This study has the potential to inform whether the Gradebook Game intervention should be adopted by other schools struggling with low student engagement; and depending on the results, it could lead to a larger, more rigorous study that would evaluate whether the Gradebook Game is effective in promoting school engagement and achievement among a diverse study population, which could be beneficial to schools and families across the nation.

ELIGIBILITY:
Inclusion Criteria:

* Student must be attending 6th grade at Alliance College-Ready Middle Academy.
* Must assent and have signed parental consent to participate.

Exclusion Criteria:

- Students whose parents are not able to provide informed consent in English or Spanish.

Ages: 7 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Participants must be 6th grade students at Alliance College-Ready Middle Academy. They need to assent and have signed parental consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Academic and Behavior Information | up to 20 times during 6 month period
  collect school grade book and behavior information weekly for 8 to 10 time points before and after the intervention is implemented.

SECONDARY OUTCOMES:
Social Emotional well being, social status and peer support | baseline and at 6 months
  Survey data will be collected via iPad using a study ID during non-content periods at school (Advisory and Enrichment). Surveys will include measures of self-reported school engagement, social-emotional well-being, and peer support.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell D Wong, MD, PhD, Study Chair — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Participants have been assigned a study ID number to link their name, address, phone number, grade book and behavior data, and survey responses. This ID will be used for all survey data collection and to identify all grade book and behavior data.
  The computer file linking the personal identifiers and the study ID number will be kept separate from the survey, grade book, and behavior data. Personally identifying information pertaining to individual participants will not be shared or made available to other researchers. Any data request will be made to the Faculty Sponsor (Mitchell Wong, MD PhD) or to the principle investigator (Ashley Lewis-Hunter, MD) and any data shared will be encrypted and will not include any personal identifying information.